CLINICAL TRIAL: NCT04838119
Title: Preoperative COVID Testing as a Predictor of Community Disease Burden
Brief Title: Preop COVID Testing Patterns
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00071985
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: Testing, preoperative
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a preoperative asymptomatic COVID screening test

SUMMARY:
This study is an investigation of preoperative asymptomatic COVID screening nationwide. The hypothesis is that because these tests are performed without reference to pretest probability of COVID-19 disease, unlike tests based on symptoms or close contact with infected individuals, these studies may represent a more unbiased sample of the local population prevalence of asymptomatic COVID disease burden.

DETAILED DESCRIPTION:
Study will gather publicly reported, aggregated statistics on positive COVID tests over time and across geographically diverse parts of the United States, summarized weekly, from the onset of the pandemic in Spring 2020 to the present time. Study will also gather contemporaneous data on weekly community COVID cases diagnosed, local positive test percentage, hospital admissions and ICU admissions for COVID-19, and deaths from COVID 19. Similar data will be obtained from a coalition of approximately 20 academic medical centers from around the United States, with Wake Forest School of Medicine, Department of Anesthesiology serving as the coordinating center. No individual patient information will be collected. Aggregated testing data, hospital disease burden, and local disease prevalence are all publicly reported.

Data will analyzed as interrupted time series.

ELIGIBILITY:
Inclusion Criteria:

* having preoperative asymptomatic COVID testing
* > or = 18 years of age

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Publicly reported aggregate data on asymptomatic preoperative COVID tests (no individual patient information)
Sampling Method: Non-Probability Sample
Enrollment: 375692 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Percentage of asymptomatic preoperative COVID-19 positive testing | March 2020-February 2021

SECONDARY OUTCOMES:
Percentage of hospitalization per geographic area | March 2020-February 2021
Percentage of death per geographic area | March 2020-February 2021
ICU census per geographic area | March 2020-February 2021
Percentage of asymptomatic preoperative COVID-19 positive testing per geographic area | March 2020-February 2021

CONTACTS AND LOCATIONS:
Overall Officials: B S Segal, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No